CLINICAL TRIAL: NCT01225874
Title: ALinC 17, Classification ©), B-precursor Induction Treatment (I)
Brief Title: Biomarkers to Classify Young Patients With Acute Lymphoblastic Leukemia (ALL) and Remission Induction Therapy in Young Patients With B-Precursor ALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9900; U10CA030969 (NIH); COG-9900 (Other: Children's Oncology Group); POG-9900 (Other: Pediatric Oncology Group); CDR0000078618 (Other: Clinical Trials.gov)
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Leukemia
Keywords: untreated childhood acute lymphoblastic leukemia; B-cell childhood acute lymphoblastic leukemia; non-T, non-B, cALLa positive, pre-B childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — calaspargase pegol; Cytarabine; Daunorubicin; Dexamethasone; Methotrexate; pegaspargase; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stratum 3 (Experimental): Patients receive oral dexamethasone twice daily on days 1-28; vincristine sulfate IV on days 1, 8, 15, and 22; pegaspargase intramuscularly (IM) on day 4, 5, or 6; cytarabine intrathecally (IT) on day 1; and methotrexate IT on day 8 (some patients also receive methotrexate IT on days 15 and 22).
  Interventions: Drug: cytarabine; Drug: dexamethasone; Drug: methotrexate; Drug: pegaspargase; Drug: vincristine sulfate
- Stratum 4 (Experimental): Patients receive oral prednisone twice daily on days 1-28; vincristine sulfate IV on days 1, 8, 15, and 22; IM SC-PEG E. coli asparaginase on days 2, 5, 8, 12, 15, and 19; daunorubicin hydrochloride IV over 15-20 minutes on days 8, 15, and 22; and methotrexate IT on days 1 and 8 (some patients also receive methotrexate IT on days 15 and 22).
  Interventions: Drug: SC-PEG E. coli L-asparaginase; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: methotrexate; Drug: prednisone

INTERVENTIONS:
Drug: SC-PEG E. coli L-asparaginase — Given IM
  Arms: Stratum 4
Drug: cytarabine — Given IT
Drug: daunorubicin hydrochloride — Given IV
  Arms: Stratum 4
Drug: dexamethasone — Given orally
  Arms: Stratum 3
Drug: methotrexate — Given IT
Drug: pegaspargase — Given IM
  Arms: Stratum 3
Drug: prednisone — Given orally
  Arms: Stratum 4
Drug: vincristine sulfate — Given IV
  Arms: Stratum 3

SUMMARY:
RATIONALE: Studying samples of blood or bone marrow from patients with cancer in the laboratory may help doctors predict how well patients will respond to treatment. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This trial is studying biomarkers to classify young patients with acute lymphoblastic leukemia (ALL) and remission induction therapy in young patients with B-precursor ALL.

DETAILED DESCRIPTION:
OBJECTIVES:

* To provide the clinical and laboratory data necessary for placing each patient with ALL onto the proper therapeutic trial. (Classification)
* To provide an administrative base to capture classification data for correlative studies in ALL treatment protocols and series of historical protocols. (Classification)
* To provide appropriate induction regimens for patients who may then enter risk specific, post-induction therapeutic trials. (Induction therapy)
* To determine the correlation between event-free survival (EFS) and the following measures of minimal-residual disease (MRD)/early response (ER): 1) the rate of peripheral blast count disappearance and the absolute blast count on day 8 as determined morphologically, by flow cytometry, and using molecular techniques; 2) Marrow morphology on day 8, and; 3) MRD as determined by flow cytometry and molecular techniques on bone marrow and peripheral blood samples on day 29. (Induction therapy)

OUTLINE: This is a multicenter study.

* Classification study: Bone marrow or peripheral blood samples are collected and may be analyzed for B- and T-lineage antigen screening; cytochemical stains; cytogenetics (karyotype); immunophenotype screening for MLL, E2A-PBX1, TEL-AML1; immunophenotype detection of minimal-residual disease (MRD); FCM ploidy (DNA index); trisomies 4 and 10 (FISH); molecular testing for BCR/ABL, MLL rearrangements, E2A-PBX1, and TEL-AML1; molecular detection of MRD - Tγ, Tδ, or IgH; acute lymphoblastic leukemia (ALL) cell bank; special T-ALL reference laboratory studies (role of tumor suppressor genes in T-ALL and drug sensitivity profiles in T-ALL); special study for mature B-ALL [t(18;14)(a24;q32)] by FISH; and hematopathology consultation concerning morphology and cytochemistry. The immunophenotype results are used to assign patients to a treatment protocol, to assign patients to post-induction (day 28) risk group and treatment for patients with B-precursor (non-T, non-B) ALL, and to use as reference laboratory MRD results.
* Induction therapy study: Patients are entered on stratum 3 (three drugs) for NCI consensus standard-risk disease (age < 10 years and WBC < 50,000/mm³) or stratum 4 (four drugs) induction therapy for NCI consensus high-risk disease (age ≥ 10 years and/or WBC ≥ 50,000/mm³ or CNS3 disease or testicular disease).

  * Stratum 3: Patients receive oral dexamethasone twice daily on days 1-28; vincristine sulfate IV on days 1, 8, 15, and 22; pegaspargase intramuscularly (IM) on day 4, 5, or 6; cytarabine intrathecally (IT) on day 1; and methotrexate IT on day 8 (some patients also receive methotrexate IT on days 15 and 22).
  * Stratum 4: Patients receive oral prednisone twice daily on days 1-28; vincristine sulfate IV on days 1, 8, 15, and 22; IM SC-PEG E. coli asparaginase IM on days 2, 5, 8, 12, 15, and 19; daunorubicin hydrochloride IV over 15-20 minutes on days 8, 15, and 22; and methotrexate IT on days 1 and 8 (some patients also receive methotrexate IT on days 15 and 22).

Based on day 29 bone marrow results, patients may start consolidation therapy, undergo retesting in a week, or receive 2 additional weeks of therapy. Additional therapy comprises oral prednisone thrice daily for 14 days; vincristine sulfate IV and daunorubicin hydrochloride IV over 15-20 minutes on days 29 and 36; and IM pegaspargase on day 29, 30, or 31. After successful remission induction, patients are assigned to COG-P9904, COG-P9905, or COG-P9906 based on the classification study.

Patients undergo bone marrow aspiration on day 8 to determine the prognostic significance of early remission in the context of this therapy.

After completion of study treatment, patients are followed up every 6 months for 4 years and annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets one of the following sets of criteria:

  * Classification study:

    * Newly diagnosed ALL*
    * Must have one of the following:

      * ≥ 25% blasts in bone marrow
      * ≥ 100,000/μl peripheral blood WBC with ≥ 75% blasts, if bone marrow aspiration is omitted for any reason other than medical contraindication
      * ≥ 30,000/μl WBC with ≥ 75% blasts, if bone marrow aspiration is omitted because of medical contraindication
    * Immunophenotype and Wright's stain morphology of blast cells consistent with acute lymphocytic leukemia
    * ≤ 21 years of age at the time of diagnosis
    * No previous registration on 9900
    * Samples must be sent for local institution and COG Reference Laboratory studies NOTE: *It is urged that a bone marrow aspiration be performed for every patient with suspected ALL. However, a marrow is not required for patients with ≥ 100,000/μl peripheral blood WBC and ≥ 75% blasts or for those patients whose clinical condition precludes performing the procedure safely. Patients with a medical contraindication to the procedure must be discussed with one of the study coordinators and must have a peripheral blood WBC of ≥ 30,000/μl with ≥ 75% blasts.
  * Induction therapy study:

    * Patients must have a confirmed diagnosis of B-precursor acute lymphoblastic leukemia
    * Patients must be 1.001 to 21.999 years at diagnosis NOTE: Patients meeting all of the above eligibility criteria are eligible for registration on 9900 whether or not they are to be entered on a COG frontline protocol for treatment of newly diagnosed ALL. Registration on 9900 is required for all legacy POG institution patients in order to be eligible for entry on the following COG ALL studies, which are either currently open or only temporarily closed: P9407, 9904, 9905, 9907, AALL0031 and AALL00P2.

PATIENT CHARACTERISTICS:

* See Disease Characteristics

PRIOR CONCURRENT THERAPY:

* Previously untreated, with the following exception:

  * Steroid treatment* in the 48-hour period just prior to study entry will be allowed provided that a physical examination and CBC with differential were performed IMMEDIATELY prior to beginning steroids and results of both are known NOTE: *Patients on chronic steroid treatment for another disease are NOT eligible for a COG New ALL protocol.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3762 (Actual)
Dates: Start 1999-12; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Collection of the clinical and laboratory data necessary for placing patients with acute lymphoblastic leukemia (ALL) onto the proper therapeutic trial (Classification)
Creation of an administrative base to capture classification data for correlative studies in ALL treatment protocols and series of historical protocols (Classification)
Creation of appropriate induction regimens for patients (Induction therapy)
Correlation between event-free survival and measures of minimal-residual disease/early response

CONTACTS AND LOCATIONS:
Overall Officials: Dale J. Pullen, MD, Study Chair — University of Mississippi Cancer Clinic

REFERENCES:
- [Derived] Escherich CS, Chen W, Li Y, Yang W, Nishii R, Li Z, Raetz EA, Devidas M, Wu G, Nichols KE, Inaba H, Pui CH, Jeha S, Camitta BM, Larsen E, Hunger SP, Loh ML, Yang JJ. Germ line genetic NBN variation and predisposition to B-cell acute lymphoblastic leukemia in children. Blood. 2024 May 30;143(22):2270-2283. doi: 10.1182/blood.2023023336. PMID 38446568